CLINICAL TRIAL: NCT06685263
Title: Development of a Perioperative Delirium Prediction Model in Patients Undergoing Cardiovascular Surgery
Brief Title: Development of Perioperative Delirium Prediction Model
Status: Not yet recruiting | Type: Observational
Sponsor: Kubra Gunes (Other)
Responsible Party: Sponsor-Investigator, Kubra Gunes, RN, MSc, Uludag University
Organization: Uludag University (Other)
Other Study IDs: 2024-15/3
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Surgery
Keywords: cardiovascular surgery; delirium; prediction model
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Development group: The development group comprises 385 individuals. Following the data collection process, the independent risk factors for the development of delirium will be identified through statistical analysis. A delirium prediction model will then be developed based on the identified risk factors.
  Interventions: Behavioral: Group 1
- Validation group: The validation group comprises 385 individuals. The delirium prediction model, constructed using the data from the development group, will be validated by testing the data from the validation group. This process will enable the evaluation of the model's suitability and calibration for predicting delirium.
  Interventions: Behavioral: Group 2

INTERVENTIONS:
Behavioral: Group 1 — The development group comprises 385 individuals. Following the data collection phase of the development group, the independent risk factors for the onset of delirium will be identified through statistical analysis. A delirium prediction model will then be constructed using the identified risk factors.
  Groups: Development group
Behavioral: Group 2 — The validation group comprises 385 individuals. The delirium prediction model created using the data from the development group will be validated by testing the data from the validation group. This will enable the evaluation of the model's fit and calibration in predicting delirium.
  Groups: Validation group

SUMMARY:
Postoperative delirium is an acute organic brain dysfunction that is commonly observed following cardiovascular surgery. It presents with acute and fluctuating changes in the level of consciousness, resulting in impaired cognitive function and perception. The incidence of delirium following cardiac surgery has been reported to range from 11.4% to 55%. In light of the challenges associated with treating delirium once it has manifested, it is imperative to prioritise the early recognition and prevention of this condition. The objective of this study was to develop a perioperative delirium risk prediction model for patients undergoing cardiovascular surgery.

DETAILED DESCRIPTION:
Postoperative delirium is associated with an increased incidence of postoperative complications, which in turn lead to cognitive dysfunction, increased mortality, and the need for long-term care. It is predicted in the literature that the early detection of delirium cases, of which 30% are known to be preventable, improves prognosis. Accordingly, a prediction model based on the identification of delirium risk factors can categorise intensive care patients into distinct risk levels according to their probability of developing delirium, thus enabling healthcare professionals to ascertain the likelihood of delirium and implement suitable preventive measures. A review of the literature reveals the existence of numerous delirium prediction models designed to identify patients at high risk of developing delirium. However, there is a paucity of studies examining models for predicting delirium risk in the context of cardiovascular surgery. The objective of this study is to develop a delirium risk prediction model for the perioperative period in patients undergoing cardiovascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Previous cardiovascular surgery
* No mental deficiency and visual and hearing impairment
* Participants' acceptance to participate in the research
* The patient is not in coma (RASS score between -3 and +4, GCS score of 10 and above)

Exclusion Criteria:

* Cardiovascular surgery under emergency conditions
* Being diagnosed with delirium, dementia, psychiatric illness and taking medication for this reason before the surgery
* Serious conditions such as cardiopulmonary resuscitation during surgery
* Alcohol and drug addiction
* Duration of mechanical ventilation exceeding 36 hours
* Dying in the intensive care unit within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to be eligible for inclusion in the study, the patient must be at least 18 years of age and must have undergone a surgical procedure on the cardiovascular system. Furthermore, the subject must not have any mental or sensory impairment, psychiatric diagnosis, or be taking medication for this purpose. Furthermore, the patient must not be in a coma, exhibit a RASS score between -3 and +4, and have a GCS score of 10 or above.
Sampling Method: Probability Sample
Enrollment: 770 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Development of a delirium risk prediction model | 1 year
  The objective of this study is to develop a perioperative delirium risk prediction model for patients undergoing cardiovascular surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nursel Vatansever, Study Director — Uludag University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudolph JL, Jones RN, Levkoff SE, Rockett C, Inouye SK, Sellke FW, Khuri SF, Lipsitz LA, Ramlawi B, Levitsky S, Marcantonio ER. Derivation and validation of a preoperative prediction rule for delirium after cardiac surgery. Circulation. 2009 Jan 20;119(2):229-36. doi: 10.1161/CIRCULATIONAHA.108.795260. Epub 2008 Dec 31. PMID 19118253
- [Background] Xu Y, Meng Y, Qian X, Wu H, Liu Y, Ji P, Chen H. Prediction model for delirium in patients with cardiovascular surgery: development and validation. J Cardiothorac Surg. 2022 Oct 1;17(1):247. doi: 10.1186/s13019-022-02005-3. PMID 36183105